CLINICAL TRIAL: NCT04149977
Title: Blood Flow Restriction Therapy in Lower Limb Extensor Injuries: A Randomized Controlled Double-Blind Study
Brief Title: Blood Flow Restriction Therapy in Lower Limb Extensor Injuries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-01269
Record Dates: First submitted 2019-10-31; First posted 2019-11-04 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Lower Limb Injury
MeSH Terms: conditions — Leg Injuries | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- blood flow restriction therapy (pressure cuff) (Experimental): The cuff will be placed around the upper thigh of the injured leg and set at a pressure that will prevent approximately 80% arterial blood flow. The machine will determine what pressure is required to reach that 80%, when placed on the leg and turned on.
  Interventions: Behavioral: Physical Therapy with pressure cuff
- blood flow restriction therapy (placebo) (Placebo Comparator): Patients with a placebo pressure will have a pressure setting, 50% lower than the effective setting as stated in the experimental arm
  Interventions: Behavioral: Physical Therapy with placebo pressure cuff

INTERVENTIONS:
Behavioral: Physical Therapy with pressure cuff — 6 weeks of physical therapy will have similar exercises to standard therapy however the patients will use a cuff around the affected leg during the exercises.
  Arms: blood flow restriction therapy (pressure cuff)
Behavioral: Physical Therapy with placebo pressure cuff — 6 weeks of physical therapy will have similar exercises to standard therapy however the patients will use a pressure cuff around the affected leg during the exercises. The pressure cuff will have 50% of the pressure that will be considered effective.
  Arms: blood flow restriction therapy (placebo)

SUMMARY:
The primary objective of the study is to determine the efficacy of blood flow restriction therapy on patients with lower limb extensor injuries by measuring pre and post blood flow restriction therapy strength and muscle mass.

DETAILED DESCRIPTION:
The purpose is to restrict venous outflow with an inflatable cuff to create a high intensity environment increases muscle hypertrophy, thus promoting a more efficient form of rehabilitation. Blood flow restriction therapy is a blood pressure cuff placed around the desired limb with a handheld device that controls the pressure exerted by the cuff. The cuff is placed around the desired limb before a specific exercise, the physical therapist determines the appropriate pressure and time, and the patient completes the exercise as they normally would. The monitor determines the limb occlusion pressure and has an automatic timer that will deflate after the specified time has elapsed. There are also audio and visual alarms that alert the user of under or over pressurization. The specific pressure will vary based on patient's tolerance and will stay consistent through each exercise. Thus far blood flow restriction therapy has been tested in patients with several pathologies but there is limited literature on its effect on lower limb extensor injuries.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age and younger than 65 years of age
* ASA class I-II
* Diagnosed with a lower limb extensor injury (quadriceps tendon rupture, patella tendon rupture, patella fracture)
* Intention to receive physical therapy as standard of care

Exclusion Criteria:

* Legally incompetent or mentally impaired (e.g. minors, Alzheimer's subjects, dementia, etc.)
* Younger than 18 years of age or older than 65
* Any patient considered a vulnerable subject
* Patients with impaired circulation, peripheral vascular compromise, previous revascularization of the extremity, or severe hypertension
* Concomitant lower extremity traumatic injuries, delaying or precluding the subject's ability to participate in the therapy
* Immobile or use of mobile assistive device prior to injury
* No prior extensor injuries
* Patients with Sickle cell anemia or venous thromboembolism
* Patients with cancer or Lymphectomies
* Patients with increased intracranial pressure
* Patients with intention to receive standard therapy and not the study therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in extensor strength of both legs | Visit 1 Day 0
  Isokinetic strength testing with a Biodex dynamometer to measure peak torque
Change in extensor strength of both legs | Visit 3 week 6
  Isokinetic strength testing with a Biodex dynamometer to measure peak torque

SECONDARY OUTCOMES:
Change in recovery, muscle strength | Visit 1 Day 0
  Having bilateral thigh circumference measured
Change in recovery, muscle strength | Visit 1 Week 6
  Having bilateral thigh circumference measured
Change in Knee function | Visit 1 Day 0
  The IKDC subjective knee evaluation form is a self-administered questionnaire which contains 18 items divided into 3 subgroups. These subgroups are symptoms, sports and daily activities and the patients current and previous levels of knee function.
Change in Knee function | Visit 3 week 6
  The IKDC subjective knee evaluation form is a self-administered questionnaire which contains 18 items divided into 3 subgroups. These subgroups are symptoms, sports and daily activities and the patients current and previous levels of knee function.

CONTACTS AND LOCATIONS:
Overall Officials: Guillem Gonzales-Lomas, MD, Principal Investigator — NYU Langone
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) may be available upon reasonable request.
  Requests should be directed to Jordan.Fried@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data.